CLINICAL TRIAL: NCT03700281
Title: Investigating the Effectiveness of a Seasonal Influenza Vaccination Promotion Campaign for Members of a Non-Profit, Community-Based Health Insurance Plan: 2018-2019
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Texas Health Science Center at Tyler (Other)
Collaborators: Sendero Health Plans, Inc. (Unknown)
Responsible Party: Principal Investigator, Eileen Nehme, Assistant Professor, The University of Texas Health Science Center at Tyler
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SenderoFlu2018
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Influenza, Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No intervention
- Messaging (Experimental): Group will be sent flu vaccine promotion messages via text, email and U.S. Mail
  Interventions: Behavioral: Messaging
- Messaging plus incentive (Experimental): Group will be sent flu vaccine promotion messages via text, email and U.S. Mail, and will be eligible to receive a gift card as incentive for receiving flu vaccine
  Interventions: Behavioral: Messaging; Behavioral: Incentive

INTERVENTIONS:
Behavioral: Messaging — The participants will receive influenza promotion emails, text messages, and U.S. mail from Sendero Health Plans.
  Arms: Messaging; Messaging plus incentive
Behavioral: Incentive — Participants will be eligible for a gift card to a local grocery store chain as an incentive for obtaining an influenza vaccine
  Arms: Messaging plus incentive

SUMMARY:
• This study will assess the effect of promotional messaging and incentives encouraging influenza vaccination in the Sendero IdealCare policy holders during the 2018-2019 Flu Season. The intervention will consist of influenza vaccination promotion/reminders from Sendero Health Plans to subscribers, including text messages, emails, and tailored direct mail outs, i.e. postcard or a personalized letter, and incentive. The study population consists of approximately 22,500 subscribers enrolled in Sendero IdealCare Plan. The intervention will last approximately four months. The primary endpoints, assessed through administrative claims data, will be getting a flu shot during the 2018-2019 season. Data collected through this study will be used to determine effective components of influenza vaccination promotion campaigns used by a health insurance plan.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in Sendero IdealCare health plan as of August 1, 2018
* Age 18 years or older

Exclusion Criteria:

* A coverage termination date listed prior to December 31, 2018.
* Sendero member records lack both a phone number and email address.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22584 (Actual)
Dates: Start 2018-10-06 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Influenza vaccination | three months
  Receipt of an influenza vaccination documented by medical or pharmacy claim.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas System Population Health, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No